CLINICAL TRIAL: NCT03249675
Title: Clinical Trial Protocol for the Evaluating a Novel Method of EEG Evoked Response Potential Analysis in Concussion Assessment, Young Adults and Adults
Brief Title: Evaluating a Novel Method of EEG Evoked Response Potential Analysis in Concussion Assessment, Young Adults and Adults
Status: Withdrawn | Type: Observational
Why Stopped: No participant were enrolled
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM 48
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Concussion, Brain
Keywords: mild Traumatic Brain Injury; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: No

GROUPS / COHORTS (2):
- ARM 1: ARM 1: Retrospective Arm: Subjects tested with BNA in the past and have been diagnosed by their physician as having Post Concussive Syndrome. Study staff will contact the subjects and obtain Informed Consent. Study physicians will then review both BNA data and Clinical data. All relevant clinical data and all available BNA data will be shared with ElMindA. Subjects may be invited for an additional BNA follow up as part of the study.
- ARM 2: ARM 2: Subjects will be prospectively enrolled in the study at the following time points when available:
  * Acute: within 2 weeks of injury
  * PCS: Subjects which sustained a concussion in the past 3 months or more, and are still experiencing symptoms related to the injury

SUMMARY:
Concussion is widely recognized as a major public health concern in the United States and worldwide. Although many concussions resolve completely and spontaneously, almost 1 in 4 patients will go on to experience post-concussion syndrome (PCS). In the United States, PCS diagnoses have increased 100% from 2010-2015. Concurrently, recent advances in EEG evoked response potential analysis have led to a novel technique for assessing brain network activation (BNA) patterns. The purpose of this study is to explore the use of BNA in individuals who are diagnosed with PCS or have the risk of experiencing PCS due to a recent injury.

DETAILED DESCRIPTION:
Mild traumatic brain injury, also known as concussion, occurs commonly in sport. The Centers for Disease Control and Prevention estimate that as many as 3.8 million sport-related concussions occur annually in the United States. Although many concussions resolve completely and spontaneously, almost 1 in 4 patients will go on to experience post-concussion syndrome (PCS). In the United States, PCS diagnoses have increased 100% from 2010-2015. Concurrently, recent advances in EEG evoked response potential analysis have led to a novel technique for assessing brain network activation (BNA) patterns. The purpose of this study is to explore the use of BNA in individuals who are diagnosed with PCS or have the risk of experiencing PCS due to a recent injury.

ElMindA, the sponsor of this study, has developed a novel method to automatically reveal functional networks of brain activity based on analysis of EEG Event Related Potential (ERP) data. This technological platform is capable of providing new metrics of brain function which can assist in patient evaluation and management. The analysis is done in two separate processes which are entirely separate and are performed independently of one another. First EEG data are recorded and analyzed from a group, or several groups, of subjects to establish a set of group patterns which characterized the brain network activity of the group. Second, EEG data from a single subject are processed to enable subject evaluation, as compared to the established group patterns. This individual analysis is the basis of the BNA scores computed for an individual subject.

Primary Objective:

• Exploratory (e.g. Hypothesis-generating) study designed to collect data that will aid in future understanding of the relationship between Post Concussion Syndrome and Electrophysiology. The results are primarily intended for scientific inquiry and development purposes.

Additional objectives:

* Exploring the relationship between the characteristics of early/acute stage Mild Traumatic Brain Injury and the subsequent development of PCS
* Collecting electrophysiological and clinical data that will serve as the basis for athlete brain health case studies.

Arm 1: Study staff will contact subjects tested in the past with BNA and were diagnosed with Post-Concussion Syndrome at their medical facility.

Arm 2: Eligible subjects treated at the study medical facility for acute concussion or Post Concussion Syndrome will be approached by the study staff.

Interested volunteers will complete a brief initial in person or phone consultation with a member of the study team and those who meet eligibility criteria and wish to participate will be invited for a study visit in the testing facility. During this visit, a member of the study team will describe the study in greater detail, verify subject eligibility, obtain informed written consent/assent for study participation, and record relevant demographic, medical history information, concussion history and clinical assessment questioners as provided by the subject or as available from subject's medical records. The subject will then have the EEG electrode cap placed on their head and will undergo the BNA test after a brief training and instructional session.

ELIGIBILITY:
Inclusion Criteria:

* Males and females Aged 12-50
* Willingness to participate in the study and the ability to give informed assent (for children) and/or consent (for the parent of a minor or adults aged 18 years of age or older for themselves).
* Subjects that are or were diagnosed with mTBI according to the standard diagnostic procedures at the investigational site in a timeframe that meets enrollment criteria.
* Subjects that are experiencing symptoms of concussion or Post-concussion Syndrome at the time of their initial test session.

Exclusion Criteria:

* Subjects that have undergone neuroimaging with identification of intracranial structural pathology.
* Self-reported history of central nervous system injury other than mTBI, or disease (examples will include, but will not be limited to, moderate or severe traumatic brain injury (TBI with a Glasgow Coma Scale < 13) epilepsy, seizures, brain surgery)
* Neuropsychological disorder such as autistic spectrum disorder
* Any history of a learning disability (examples include, but will not be limited to, dyslexia, dysgraphia, dyscalculia, or a nonverbal learning disorder)
* Use of any medication affecting central nervous system (CNS) in the past 3 months prior to their BNA (i.e. antidepressants, anticonvulsants, psychostimulants, first generation antihistamines, etc.)
* Active head lice infection
* Open scalp wound
* baldness, dread locks or hair that is otherwise sufficiently long and thick so as to preclude appropriate scalp electrode cap fit
* Deafness, and/or blindness

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents, young adults and adults of both genders.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Developing a BNA database for concuss population. | This study duration is 18 months
  Functional networks of brain activity in healthy individuals measured using analysis of EEG Event Related Potential (ERP) data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kutcher, MD, Principal Investigator
Locations (1):
- The Sports Neurology Clinic at The CORE Institute, Brighton, Michigan, United States